CLINICAL TRIAL: NCT02313181
Title: Early Limited Formula for Treating Lactation Concerns
Acronym: ELF-TLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Milton S. Hershey Medical Center (Other); HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Valerie Flaherman, Associate Professor of Pediatrics and Epidemiology and Biostatistics, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R40-MC26810
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Breastfeeding
Keywords: breastfeeding; lactation; newborn
MeSH Terms: conditions — Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Limited Formula (Experimental): 10 milliliters (mL) Nutramigen fed to baby by syringe after each breastfeeding and discontinued at the start of mature milk production
  Interventions: Other: Early Limited Formula
- Standard Care (Other): Continue exclusive breastfeeding unless otherwise instructed by a health care provider
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Early Limited Formula — 10 milliliters (mL) Nutramigen fed to baby by syringe after each breastfeeding and discontinued at the start of mature milk production
  Other Names: ELF
  Arms: Early Limited Formula
Other: Standard Care — Continue exclusive breastfeeding unless otherwise directed by a health care provider
  Arms: Standard Care

SUMMARY:
This is a randomized, controlled trial designed to evaluate a new strategy for promoting continued breastfeeding for mothers and babies who initiated breastfeeding in the newborn period. The new strategy, called Early Limited Formula (ELF), consists of 10mL of formula fed to each baby by syringe after each breastfeeding prior to the onset of mature milk production. The study intervention is discontinued at the onset of mature milk production, and the investigators will then follow mothers and infants for 12 months to assess the effect of ELF on breastfeeding duration, maternal experience and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Full term, healthy singleton infant (≥ 37 0/7 weeks gestational age) in well newborn nursery
2. Exclusively breastfeeding (has not received any feedings other than breast milk)
3. Infant is 18-72 hours old
4. Infant has weight loss of ≥75th percentile on delivery mode specific nomogram documented at 12-72 hours of age
5. English-speaking mother

Exclusion Criteria:

1. Mothers or infants for whom breastfeeding is not recommended by the clinical team
2. Mothers who have already begun to produce mature breast milk
3. Any formula or water feeding prior to enrollment
4. Infants who have already lost ≥10% of their birth weight
5. Family with no active telephone number (home or cellular)
6. Plan for infant adoption or foster care
7. Mothers <18 years of age
8. Infant receiving scoring for Narcotic Abstinence Syndrome -

Ages: 18 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 328 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Length of breastfeeding duration | 12 months
  The investigators will follow babies for 12 months to determine how long the babies continued breastfeeding

SECONDARY OUTCOMES:
State Trait Anxiety Inventory | 1 month
  The investigators will follow mothers for 1 month to measure their responses on the State Trait Anxiety Inventory.
Health care utilization | 1 month
  The investigators will follow babies for 1 month to determine how often they were seen by an outpatient provider, inpatient provider or emergency provider.
Formula use | 6 months
  The investigators will follow babies for 6 months to determine the volume of formula used.

OTHER OUTCOMES:
Edinburg Postnatal Depression Scale | 1 month
  The investigators will follow mothers for 1 month to determine their score on the Edinburg Postnatal Depression Scale
Breastfeeding Self-Efficacy Scale | 1 month
  The investigators will follow mothers for 1 month to determine their score on the Breastfeeding Self-Efficacy Scale
Satisfaction with Quality of Care | 1 month
  The investigators will follow mothers for 1 month to determine their score on the Satisfaction with Health Care Following Childbirth Scale
Milk supply concern | 1 month
  The investigators will follow mothers for 1 month to determine their score on the Infant Satisfaction and Satiety Subscale

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flaherman, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco Medical Center, San Francisco, California
  - Penn State Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Derived] Flaherman VJ, Cabana MD, McCulloch CE, Paul IM. Effect of Early Limited Formula on Breastfeeding Duration in the First Year of Life: A Randomized Clinical Trial. JAMA Pediatr. 2019 Aug 1;173(8):729-735. doi: 10.1001/jamapediatrics.2019.1424. PMID 31157878
- [Derived] Flaherman VJ, Narayan NR, Hartigan-O'Connor D, Cabana MD, McCulloch CE, Paul IM. The Effect of Early Limited Formula on Breastfeeding, Readmission, and Intestinal Microbiota: A Randomized Clinical Trial. J Pediatr. 2018 May;196:84-90.e1. doi: 10.1016/j.jpeds.2017.12.073. Epub 2018 Mar 14. PMID 29550235